CLINICAL TRIAL: NCT06996392
Title: Phase I Trial of QH-1A Hybrid Bio-Artificial Liver With Ex Vivo Blood-Purifying MSCs in Acute-on-Chronic Liver Failure: Safety, Efficacy, and Treatment Schedule Exploration
Brief Title: Phase I Trial of QH-1A Hybrid Bio-Artificial Liver With Ex Vivo Blood-Purifying MSCs in Acute-on-Chronic Liver Failure
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Guangdong Qianhui Biotechnology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Liang Peng, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PL20
Record Dates: First submitted 2025-05-11; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: Acute -On-Chronic Liver Failure; Bio-artificial liver; Mesenchymal stem cells
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 4-hour group (Experimental): The 4-hour group will receive a single biological artificial liver treatment for 4 hours (±15 minutes).
  Interventions: Combination Product: Combining the QH-1A bioartificial liver device with mesenchymal stem cells for blood purification（4 hours）
- 6-hour group (Experimental): The 6-hour group will receive a single biological artificial liver treatment for 6 hours (±15 minutes).
  Interventions: Combination Product: Combining the QH-1A bioartificial liver device with mesenchymal stem cells for blood purification（6 hours）
- 8-hour group (Experimental): The 8-hour group will receive a single biological artificial liver treatment for 8 hours (±15 minutes).
  Interventions: Combination Product: Combining the QH-1A bioartificial liver device with mesenchymal stem cells for blood purification（8 hours）
- Multiple-treatment group (Experimental): The Safety Evaluation Committee will determine the maximum tolerable treatment duration based on the 28-day safety observation outcomes from the 4-, 6-, and 8-hour groups. This duration will then be adopted as the treatment time for the multiple-treatment group. Subjects in the multiple-treatment group will undergo 2-3 treatments at this maximum duration, with an interval of 3 (±1) days between sessions.
  Interventions: Combination Product: Combining the QH-1A bioartificial liver device with mesenchymal stem cells for blood purification（Multiple-treatment）

INTERVENTIONS:
Combination Product: Combining the QH-1A bioartificial liver device with mesenchymal stem cells for blood purification（4 hours） — The 4-hour group treatment session lasts 4 hours (±15 minutes). In the HBAL mode of the combined bioartificial liver device QH-1A, blood is initially filtered to separate the plasma, which is then pumped into a bioreactor. In this study, this bioreactor is uniquely filled with immortalized mesenchymal stem cells (PT-MSCs) optimized for blood purification. These cells are cultured to adhere to the outer surface of hollow fibers within the bioreactor, creating a stable and efficient living interface that continuously secretes bioactive factors such as exosomes.After passing through the bioreactor, the plasma is re-filtered and then returned to the patient's circulation via a dedicated pump.
  Arms: 4-hour group
Combination Product: Combining the QH-1A bioartificial liver device with mesenchymal stem cells for blood purification（6 hours） — After the three subjects in the 4-hour group completed their 4-week follow-up, the Safety Evaluation Committee convened a meeting to review the safety data and determine whether to proceed with the recruitment for the 6-hour group.The 6-hour group treatment session lasts 6 hours (±15 minutes).The treatment procedure is identical to that of the 4-hour group.
  Arms: 6-hour group
Combination Product: Combining the QH-1A bioartificial liver device with mesenchymal stem cells for blood purification（8 hours） — After the three subjects in the 6-hour group completed their 4-week follow-up, the Safety Evaluation Committee convened a meeting to review the safety data and determine whether to proceed with the recruitment for the 8-hour group. The 8-hour group treatment session lasts 8 hours (±15 minutes).The treatment procedure is identical to that of the 4-hour group.
  Arms: 8-hour group
Combination Product: Combining the QH-1A bioartificial liver device with mesenchymal stem cells for blood purification（Multiple-treatment） — Subjects in the multiple-treatment group will receive 2-3 sessions of bioartificial liver treatment; the number of sessions will be determined by the investigators based on the subjects' clinical needs. The treatment duration for each session will be set as the maximum tolerable period, as confirmed by the Safety Evaluation Committee based on 28-day safety observations from the 4-hour, 6-hour, and 8-hour groups. Each treatment session is administered following the procedure applied to patients in the group with the optimal tolerability duration.
  Arms: Multiple-treatment group

SUMMARY:
The goal of this Phase I clinical trial is to evaluate the safety and efficacy of combining the QH-1A bioartificial liver device with mesenchymal stem cells（MSCs） for blood purification in treating patients with acute-on-chronic liver failure, and to determine the optimal treatment duration and frequency for Phase II. The study will enroll patients aged 18 to 65 years who meet the diagnostic criteria for acute-on-chronic liver failure as outlined in the 2024 Chinese Liver Failure Clinical Guidelines.

The main questions this study aims to answer are:

* Does the combined therapy improve the 28-day survival rate after the final treatment?
* Does the QH-1A device in its HBAL mode consistently achieve the predefined device performance pass rate?
* Do patients show significant improvements in their biochemical markers following treatment?
* What is the immunogenicity profile of the mesenchymal stem cells used for blood purification?

Participants will be screened within 14 days before their first treatment and will be allocated into one of four groups based on treatment duration and frequency:

* 4-hour group (3 patients)
* 6-hour group (3 patients)
* 8-hour group (3 patients)
* Multiple-treatment group (6 patients) Treatment will be administered in a sequential escalation-from the 4-hour group up to the multiple-treatment group-based on safety data from a 28-day observation period, which will be reviewed by a Safety Evaluation Committee. In addition, upon referral to the Hepatitis B Health Clinic, participants will receive tailored health education, comprehensive liver function and virological assessments, and an individualized treatment and follow-up plan.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years, irrespective of gender.
* Patients with acute-on-chronic liver failure, diagnosed according to the - - Guideline for diagnosis and treatment of liver failure (2024 version) in China.
* Subjects must provide informed consent prior to the study and voluntarily sign the written informed consent form.
* Subjects must be able to communicate effectively with the investigators and comply with the study protocol.

Exclusion Criteria:

* Active bleeding or disseminated intravascular coagulation (DIC) that is not effectively controlled.
* Allergies to the blood products or medications used during treatment.
* Circulatory failure.
* Occurrence of myocardial infarction, cerebral infarction, or cerebral hemorrhage within the past 6 months.
* A history of malignant tumors within the past 5 years (except for cured basal cell carcinoma of the skin or carcinoma in situ of the cervix).
* Any other conditions that, in the opinion of the investigator, render the subject unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 28-day

SECONDARY OUTCOMES:
Combined Bioartificial Liver Device QH-1A Equipment Performance Pass Rate | Day 1
  Pass Criteria: If all items on the trial medical device evaluation are rated as "Yes," the device's performance is deemed acceptable. If any evaluation item is rated as "No," the device's performance is considered unacceptable. Reasons for any "No" ratings must be documented.
Changes from the baseline in Child-Pugh grade | 28-day
  The Child-Pugh classification evaluation indicators consist of hepatic encephalopathy, ascites, total bilirubin, albumin, and prolonged PT time. The scoring and classification of the severity of Child-Pugh liver diseases are as follows:Grade A is 5 to 6 points. Grade B is 7 to 9 points. Grade C is 10 to 15 points. The higher the score, the worse the liver function.
Changes from the baseline in COSSH-ACLF IIs | 28-day
  The Chinese Severe Hepatitis B Study Group (COSSH), based on a multicenter, open-label large cohort study, has established a novel prognostic scoring system for hepatitis B virus (HBV)-ACLF: COSSH-ACLF II s. A score of less than 7.4 indicates a low-risk group, a score between 7.4 and 8.4 indicates a moderate-risk group, and a score greater than 8.4 indicates a high risk of 28- and 90-day mortality.
Changes from the baseline in MELD score | 28-day
  The MELD score (Model for End-Stage Liver Disease) is a scoring system used to assess the urgency of liver transplantation in chronic liver disease patients. The MELD score typically ranges from 6 to 40, with higher scores indicating more severe disease and a greater need for liver transplantation.
The rate of bridging liver transplantation | 28-day

OTHER OUTCOMES:
Incidence of adverse events and serious adverse events | 28-day
  All treatment-related adverse events will be assessed by CTCAE v5.0.
Number of participants with positive infectious pathogens in the return fluid | Day1
  After each treatment session (0-15 minutes post-treatment), the return fluid from the bioreactor will be collected for testing of infectious pathogens (bacteria, fungi) and endotoxins.
Number of participants with positive replicative lentivirus in the blood | Day1,Day28
  blood samples were collected for the detection of replicative lentivirus.
Number of participants in whom mesenchymal stem cell shedding was detected in the return fluid | Day1
  During each treatment process, return fluid is collected at the front and back of the reactor at designated time points. Techniques such as flow cytometry and real-time fluorescence quantitative PCR are used to assess the shedding of mesenchymal stem cells.
Changes from the baseline in immunogenicity indicators | Day1, Day7,Day28
  During the observational study, changes in immunogenicity indicators were monitored to evaluate the immunogenicity of the investigational product. The immunogenicity indicators included immunoglobulins (IgM, IgG, IgA, IgE), complements (C3, C4), lymphocyte subset analysis (CD3+ T cell count and percentage, CD4+ T cell count and percentage, CD8+ T cell count and percentage), and cytokines (IL-2, IL-6, IL-8, IL-10, TNF-α, IFN-γ).
  Blood samples were collected for immunogenicity assessment at the following time points: before each machine-based treatment (-30 min to 0 min), 7±1 days, 28±3 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No